CLINICAL TRIAL: NCT00171600
Title: Comparative, Open Multicenter Trial Assessing the Effect on Albumin Excretion Rate of 320mg Valsartan (With or Without HCTZ) vs 40mg Lisinopril (With or Without HCTZ) on Hypertensive Patients With Diabetic and Non-diabetic Nephropathy and Albuminuria
Brief Title: Antialbuminuric Effects of Valsartan and Lisinopril
Status: Terminated | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CVAL489AES15
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Last update posted 2011-11-08 (Estimated); Status verified 2011-11

CONDITIONS: Hypertension; Early Diabetic Nephropathy
Keywords: valsartan; lisinopril; albuminuria; diabetic nephropathy
MeSH Terms: conditions — Hypertension; Diabetic Nephropathies; Albuminuria | interventions — Valsartan; Hydrochlorothiazide; Lisinopril

INTERVENTIONS:
Drug: VALSARTAN, VALSARTAN PLUS HCTZ, LISINOPRIL, LISINOPRIL PLUS HCTZ

SUMMARY:
Title: Antialbuminuric effect of valsartan, lisinopril and valsartan versus lisinopril in non-diabetic and diabetic renal disease: a randomized (3:3:1), open label, parallel group, 20 weeks follow-up.

Objective: To evaluate the antialbuminuric effect of high doses of valsartan vs lisinopril vs combo treatment in non-diabetic and diabetic patients.

Hypothesis: Combo treatment reduces microalbuminuria and the albumin/creatinine ratio more than monotherapies..

Design: Multicentric, randomized, open label, parallel group, active controlled.

Dose / regimen: Valsartan 320 vs Lisinopril 40 vs Valsartan/lisinopril 160/20

Primary Endpoint: Antialbuminuric effect of valsartan 320 mg, lisinopril and valsartan versus lisinopril 40 mg in non-diabetic and diabetic renal disease following 5 months of follow-up. Description % of change in albuminuria from baseline at 20 weeks.

Secondary Endpoint : To investigate the effect of 5 months treatment with valsartan,lisinopril and valsartan versus lisinopril in GFR (Cl creatinine), also to investigate the effect of 5 months treatment with valsartan, lisinopril and valsartan plus lisinopril on blood pressure and the effect on left ventricular mass index using electrocardiogram and Cornell-Sokolow method.

ELIGIBILITY:
Inclusion Criteria:

* Male or female outpatients aged 40-75 years,
* Chronic nephropathy, as defined by a serum creatinine concentration of > 1.3 mg/dL or calculated glomerular filtration rate of > 30 mL/min/1.73 m2.
* Persistent albuminuria, as defined by urinary albumin excretion exceeding 20 mg/ 24 h but not > 1000 mg/ 24h. (for a minimum of three months).
* Hypertensive patients not adequately controlled with or without treatment (controlled: <130/80 mmHg).
* Written informed consent to participate in the study prior to any study procedures.

Exclusion Criteria:

* Immediate need for renal replacement therapy.
* Treatment resistant oedema or nephrotic syndrome.
* Need for treatment with corticosteroids, non-steroidal antiinflammatory drugs, or immunosuppressive drugs.
* Albuminuria greater than 1000mg /24h and or less than 20mg/24h.
* Total cholesterol < 135mg/dl or not need for statins treatment.
* Renovascular hypertension
* Malignant hypertension
* MI, cerebrovascular accident within last year, severe peripheral vascular disease, CHF, chronic hepatic disease.
* Angiotensin converting enzyme inhibitors and angiotensin II receptors blockers within one month prior to randomization.
* A serum creatinine concentration >265 umol/L

Ages: 40 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2005-07; Primary Completion 2007-01 (Actual); Study Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
Change from baseline in urine albumin excretion rate from collected urine samples, after 16 and 20 weeks

SECONDARY OUTCOMES:
Blood pressure less than 130/80 mmHg after 16 and 20 weeks of treatment
Change from baseline 48-hour ambulatory blood pressure, and blood pressure less than 130/80 mmHg after 16 and 20 weeks of treatment
Blood pressure less than 130/80 mmHg at night, measured by 48-hour ambulatory blood pressure monitoring, after 16 and 20 weeks of treatment
Change from baseline in size of left heart ventricle by electrocardiogram (ECG) after 20 weeks
Change from baseline in kidney function after 16 and 20 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis Pharmaceuticals, Basel, Switzerland

REFERENCES:
- [Derived] Natale P, Palmer SC, Navaneethan SD, Craig JC, Strippoli GF. Angiotensin-converting-enzyme inhibitors and angiotensin receptor blockers for preventing the progression of diabetic kidney disease. Cochrane Database Syst Rev. 2024 Apr 29;4(4):CD006257. doi: 10.1002/14651858.CD006257.pub2. PMID 38682786